**Study:** A Feasibility Study of Integrating Maternal, Infant and Young Child Nutrition (MIYCN) Counselling Services in Urban Maternal, Neonatal and Child Health (MNCH)

Services in Bangladesh: A Quasi-experimental Evaluation

Clinicaltrials.gov: NCT03882268

**Document date:** August 6, 2021

# Written informed consent form for service providers, supervisors and managers of the service providers

**Protocol Title:** A Feasibility Study of Integrating Maternal, Infant and Young Child Nutrition (MIYCN) Counselling Services in Urban Maternal, Neonatal and Child Health (MNCH) Services in

Bangladesh: A Quasi-experimental Evaluation

Principle Investigator's name: Dr. Phuong Hong Nguyen

**Organization:** The research project carried out by the International Food Policy Research Institute (IFPRI), USA and Data Analysis and Technical Assistant Limited (DATA), Bangladesh

## **Purpose of the research:**

We work at the International Food Policy Research Institute (IFPRI) and Data Analysis and Technical Assistant Limited (DATA). We are collecting information to study how MIYCN counselling services can be integrated into MNCH services in urban centres in Dhaka. The aim of this study is to evaluate how integrating these services can improve service delivery and drive behaviour change. The understanding gained from this study will be utilized for planning better National Nutrition Services in Bangladesh as well as in your community.

#### Why have we selected you?

Since you are providing different nutrition services through your regular service delivery during antenatal (ANC) and child contacts (both well child for immunization and sick child contacts) at this facility, we are inviting you to participate in this study.

# What is expected from the respondent?

If you agree to participate in the study we would like to ask you questions regarding your workload, supervision, training, and other factors related to your service delivery. The interview will last approximately 30-40 minutes. We would also like to observe the antenatal check-up session or immunization, or sick child visit or counselling services provided by you. We will also seek permission from your client prior to observing the procedures.

In addition, we would perform a facility assessment, using observation checklists to understand the services provided and the facilities at the clinic. In course of health facility assessment, we would require your assistance in filling up the observation checklist. We would like to use the information from this study for further improvement of services at this facility and others like it. This and any other information we observe will only be shared among the researchers in the team.

Please rest assured that if you like to withdraw from the study at any point, you may do so without any restrictions from the investigators. Refusal to participate in the study will not cause you any harm.

#### **Risks:**

Contact with our survey team presents a risk of spreading COVID-19, an illness that can spread from person to person. To protect you, our survey team members will maintain two meters of distance, wear a mask, and wash or sanitize hands before and after the interview. We will also provide you with a mask. Each member of our survey team was checked for any symptoms of COVID-19 before starting work today. We ask that you let us know whether you have experienced any COVID-19 related symptoms today, so that additional safety measures can be applied if needed.

There will be no other risks related to your participation in this study. The observation will only be based on the regular activities you perform for antenatal services or management of child visits. During the interview, you will be asked questions on your workload, knowledge, motivation and service provision. You have the right to not allow us to observe if you are uncomfortable with any of the activities you perform.

#### **Benefits:**

Participation in this study may not benefit you directly. However, it gives you an opportunity to get evaluated on your activities regarding antenatal check-up and child visits which will contribute in improving quality of nutritional services that you deliver to your community.

#### Privacy, anonymity and confidentiality:

We do hereby affirm that privacy, anonymity and confidentiality of information identifying you will strictly be maintained. None other than the investigators of this research, legal and ethical authorities would have access to the information. We would not use or record your name rather we will use a unique code so all information is kept confidential.

#### **Future use of information:**

Anonymous information and data may be presented only for the stated objectives of the study. We, in no circumstance, will use your name or contact address. Your provided information might be used in publications, presentations or in developing government documents. However, this will not conflict with or violate the maintenance of privacy, anonymity and confidentiality of information identifying participants in any way.

#### Right not to participate and withdraw:

Your participation in the study is voluntary, and you have the sole authority to decide for or against your participation. You do not have to comply with the selected procedure that you do not want to. You would also be able to withdraw from participation any time during the study, without showing any cause. Refusal to participate in the study will not cause you any harm or change the benefits that you used to receive from this facility.

#### **Principle of compensation:**

As mentioned earlier, your participation in this study is completely voluntary and you will not get any payment for participating in this study.

## **Contact person:**

If you have questions about this study or if you feel that you have been treated unfairly or have been hurt by joining the study, you may communicate with the Principal Investigator of the study Dr. Phuong Hong Nguyen at <u>p.h.nguyen@cgiar.org</u> or Dr. Md. Zahidul Hassan at hassanzahidul@gmail.com, phone number 01711535999.

If you agree to our proposal of enrolling in our study, please indicate that by putting your signature at the specified space below. Thank you for your cooperation

#### **Participant's statement:**

My signature below indicates that I have understood the contents and objectives of the study and the associated risk or benefits and I have received answers to all of my queries. I am voluntarily participating in the study and I have been told who to contact with if I have any question or complaint. I am aware that I will be given a copy of this consent form for my own records.

| Signature of participant | Date |
|---|---|
| Witness: I certify that all the above inform he/she understood the explanation. | nation was adequately explained to the participant and |
| Signature or of the witness | Date |

# Written informed consent form for clients

**Protocol Title:** A Feasibility Study of Integrating Maternal, Infant and Young Child Nutrition (MIYCN) Counselling Services in Urban Maternal, Neonatal and Child Health (MNCH) Services in

Bangladesh: A Quasi-experimental Evaluation

Principle Investigator's name: Dr. Phuong Hong Nguyen

**Organization:** The research project carried out by the International Food Policy Research Institute (IFPRI), USA and Data Analysis and Technical Assistant Limited (DATA), Bangladesh

#### **Purpose of the research:**

We work at the International Food Policy Research Institute (IFPRI) and Data Analysis and Technical Assistant Limited (DATA). We are collecting information to study how MIYCN counselling services can be integrated into MNCH services in urban centres in Dhaka. The aim of this study is to evaluate how integrating these services can improve service delivery and drive behaviour change. The understanding gained from interviews with clients as well as direct observation of service delivery will be utilized for planning better National Nutrition Services in Bangladesh as well as in your community.

#### Why we have selected you?

Since you have received health care services for yourself or your child from this health facility, we want to know about your experience of receiving the service and type of nutritional services and messages you received from health care providers, and to observe your visit with your provider. Therefore, we are inviting you to participate in this study.

#### What is expected from the respondent?

If you agree to participate in the study we would like to interview you prior to your ANC/child visit, observe your session with your provider, and ask you some brief questions about your satisfaction with services after your session. The segment of the interview prior to your healthcare visit will last 30-40 minutes, and the post-session interview will last 5-10 minutes. We would like to use the information from this study for further improvement of the nutritional health services. This and any other information we observe will only be shared among the researchers in the team.

Please rest assured that if you like to withdraw from the study at any point, you may do so without any restrictions from the investigators. Refusal to participate in the study will not cause you any harm.

## Risks:

Contact with our survey team presents a risk of spreading COVID-19, an illness that can spread from person to person. To protect you, our survey team members will maintain two meters of distance, wear a mask, and wash or sanitize hands before and after the interview. We will also provide you with a mask. Each member of our survey team was checked for any symptoms of COVID-19 before starting work today. We ask that you let us know whether you have experienced any COVID-19 related symptoms today, so that additional safety measures can be applied if needed.

There will be no other risks related to your participation in this study. The observation will only be based on the regular services you receive during your ANC or child visit. Similarly, questions you are asked will be based on services you received today and in the past at this facility, and your satisfaction with the care you received. You have the right to not allow us to observe if you are uncomfortable at any time.

#### **Benefits:**

Participation in this study may not benefit you directly, but the results of the study may be used to improve the services that you and others in your community receive.

#### Privacy, anonymity and confidentiality:

We do hereby affirm that privacy, anonymity and confidentiality of information identifying you will strictly be maintained. None other than the investigators of this research, legal and ethical authorities would have access to the information. We would not use or record your name rather we will use a unique code so all information is kept confidential.

#### **Future use of information:**

Anonymous information and data may be presented only for the stated objectives of the study. We, in no circumstance, will use your name or contact address. Your provided information might be used in publications, presentations or in developing government documents. However, this will not conflict with or violate the maintenance of privacy, anonymity and confidentiality of information identifying participants in any way.

## Right not to participate and withdraw:

Your participation in the study is voluntary, and you have the sole authority to decide for or against your participation. You do not have to comply with the selected procedure that you do not want to. You would also be able to withdraw from participation any time during the study, without showing any cause. Refusal to participate in the study will not cause you any harm or change the benefits that you used to receive from this facility.

# **Principle of compensation:**

As mentioned earlier, your participation in this study is completely voluntary and you will not get any payment for participating in this study.

#### **Contact person:**

If you have questions about this study or if you feel that you have been treated unfairly or have been hurt by joining the study, you may communicate with the Principal Investigator of the study Dr. Phuong Hong Nguyen at <a href="mailto:p.h.nguyen@cgiar.org">p.h.nguyen@cgiar.org</a> or Dr. Md. Zahidul Hassan at <a href="mailto:hassanzahidul@gmail.com">hassanzahidul@gmail.com</a>, phone number 01711535999.

If you agree to our proposal of enrolling in our study, please indicate that by putting your signature at the specified space below. Thank you for your cooperation

## **Participant's statement:**

My signature below indicates that I have understood the contents and objectives of the study and the associated risk or benefits and I have received answers to all of my queries. I am voluntarily participating in the study and I have been told who to contact with if I have any question or complaint. I am aware that I will be given a copy of this consent form for my own records.

| Signature of participant | Date | |
|---|---|---|
| Witness: I certify that all the above informulae/she understood the explanation. | nation was adequately explained to the participant | t and |
| Signature or of the witness | Date | |